CLINICAL TRIAL: NCT03766529
Title: Loop Isolation-based Uploading Pre-conditioning to Protect Heart From Ischemic-Reperfusion Damage in Coronary Artery Bypass Surgery
Brief Title: Loop Isolation-based Uploading Pre-conditioning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Clinical Investigator, Nanjing Medical University
Other Study IDs: LiuPhD
Record Dates: First submitted 2018-12-03; First posted 2018-12-06 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Ischaemic Heart Diseases
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: loop isolation-based uploading preconditioning (LiuPhD) — declamping was not done until heart could resume normal mechanical activities and sustain well for three minutes in terms of heart rate, rhythm, and myocardial contractility via continuous antegrade warm blood delivery closely following TWBC reperfusion.

SUMMARY:
Myocardial protection is of crucial importance for surgical coronary revascularization in patients with ischaemic heart diseases. The investigators proposed loop isolation-based uploading preconditioning to protect heart from ischemic-reperfusion damage (LiuPhD) as a novel cardioprotective strategy, and applied to patients who underwent on-pump coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
Myocardial protection is of crucial importance for surgical coronary revascularization in patients with ischaemic heart diseases. Considerable effort has been made to optimize cardioprotective strategy for improving cardiac performances after global myocardial ischemia. Of various strategies, terminal warm blood cardioplegia (TWBC) delivery has been proven to be effective in reducing risk of ischemic attack at the time of myocardial reperfusion. Based on TWBC strategy and Frank-Starling law of heart, the investigators proposed loop isolation-based uploading preconditioning to protect heart from ischemic-reperfusion damage (LiuPhD) as a novel myocardial protective strategy, which procedurally renders coronary loop via brief warm blood delivery independent of extracorporeal loop following TWBC delivery just before declamping. The investigators hypothesize that LiuPhD strategy allows myocardial cells complete depolarization and drives heart into zero-loading heat cycles, contributing to enhancing myocardial physiologic reserve and improving cardiac initiative capacity responding to upcoming loading increases after onset of clamp release. The aim of the present study was to determine whether LiuPhD strategy during on-pump coronary artery bypass grafting (CABG) can attenuate reperfusion injury after global myocardial ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a first, elective, isolated, open thoracotomy, on-pump CABG were eligible for enrollment if they if they had coronary angiography-confirmed unprotected left main disease, 3-vessel disease with or without proximal LAD artery disease, or 2-vessel disease with proximal LAD artery disease.
* Inclusion criteria were evidence of preserved left ventricular function (LVEF≥35%) and normal or mild pulmonary hypertension (sPAP<50mmHg).

Exclusion Criteria:

* Exclusion criteria were secondary CABG, emergency CABG, conversion operations form off-pump CABG or minimally invasive CABG surgery, or any additional cardiac lesions necessitating concomitant surgery, as well as being considered too high risk for surgical revascularization.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The LiuPhD (Loop Isolation-based Uploading Preconditioning to Protect Heart from ischemic-reperfusion Damage) study was a prospective, open-label, single-arm, first-in-man trial on the use of LiuPhD strategy for myocardial protection in patients who underwent surgical coronary revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of postoperative maximum cardiac troponin T | up to 30 days
  postoperative maximum concentration serum cardiac troponin T (cTnT) as markers of myocardial injury.

CONTACTS AND LOCATIONS:
Locations (1):
- TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided